CLINICAL TRIAL: NCT05550636
Title: The Effect of Multiple Oral Doses of BI 1015550 on Metabolism of Midazolam Administered Orally in Healthy Male Subjects (Open-label, Two-period Fixed Sequence Design Trial)
Brief Title: A Study in Healthy Men to Test Whether BI 1015550 Influences the Amount of Midazolam in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0033; 2022-002249-16 (EudraCT Number)
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 1015550 + midazolam treatment arm (Experimental): test and reference treatment arm
  Interventions: Drug: BI 1015550; Drug: midazolam

INTERVENTIONS:
Drug: BI 1015550 — BI 1015550
  Other Names: Nerandomilast; JASCAYD®
Drug: midazolam — midazolam

SUMMARY:
The main objective of this trial is to investigate the induction effect of multiple doses of BI 1015550 on the pharmacokinetics of the sensitive CYP3A4 substrate midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, two period fixed sequence design trial to investigate the induction effect of multiple oral doses of 18 milligram (mg) of BI 1015550 twice daily (bid) on the pharmacokinetics of a single oral dose of midazolam.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to treatment if any of the entry criteria were violated.
Groups:
- Midazolam (R) / BI 1015550 + Midazolam (T): A single dose of 1 milliliter (mL) of midazolam solution (2mg/mL) was administered orally on Day 1 as reference treatment (R ) in period 1. In period 2, one film-coated tablet of 18 mg BI 1015550 was administered orally twice daily (bid) for 13 days (Day -13 to Day -1), and once daily (qd) on Day 1 together with a single dose of 1 mL oral solution of midazolam (2mg/mL) as test treatment (T). There was a washout period of at least 24 hours between the reference treatment (R) and the first BI 1015550 administration in the test treatment (T).
Period: Period 1 (Reference treatment period)
Arm/Group | Midazolam (R) / BI 1015550 + Midazolam (T)
Started | 15
Completed (Completed treatment in period 1) | 15
Not Completed | 0
Period: Period 2 (Test treatment period)
Arm/Group | Midazolam (R) / BI 1015550 + Midazolam (T)
Started | 15
Completed (Completed treatment in period 2) | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all subjects who were treated with at least 1 dose of trial drug.
Arm/Group | Midazolam (R) / BI 1015550 + Midazolam (T)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of midazolam in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  Detailed timeframe:
  For midazolam (R): Within 3 hours prior to midazolam administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after midazolam administration in period 1.
  For BI + midazolam (T): 313 hours prior to administration of BI 1015550 + midazolam, at BI 1015550 + midazolam administration (0 hour) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after administration of BI 1015550 + midazolam in period 2.
Time Frame: Midazolam (R): Within 3 hours prior to midazolam administration and up to 24 hours after midazolam administration, in period 1. BI 101550 + midazolam (T): 313 hours prior and up to 24 hours after BI 1015550 + midazolam administration, in period 2.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): this set included all subjects in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: Hours * nanomol per liter (h*nmol/L)
Groups:
- Midazolam (R): A single dose of 1 mL of midazolam solution (2mg/mL) was administered orally on Day 1 as reference treatment (R ) in period 1.
- BI 1015550 + Midazolam (T): One film-coated tablet of 18 mg BI 1015550 was administered orally twice daily (bid) for 13 days (Day -13 to Day -1), and once daily (qd) on Day 1 together with a single dose of 1 mL oral solution of midazolam (2mg/mL) as test treatment (T) in period 2.
Arm/Group | Midazolam (R) | BI 1015550 + Midazolam (T)
Number analyzed (Participants) | 15 | 15
Hours * nanomol per liter (h*nmol/L) | 75.1 (NA) — Adjusted geometric standard error (gSE) = 1.108 | 69.3 (NA) — Adjusted geometric standard error (gSE) = 1.108
Statistical Analysis 1: Comparison: Midazolam (R) vs BI 1015550 + Midazolam (T); The statistical model used was an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoint was logtransformed (natural logarithm) prior to fitting the ANOVA model. This model includes effects accounting for the sources of variation: treatment. The effect 'subjects' is considered as random, whereas the treatment effect is considered as fixed. Quantities were then back-transformed to the original scale to provide the point estimate and 90% confidence interval; Test type: Other; adjusted gMean Ratio (%) = 92.3, 90% CI 2-sided [79.3 to 107.4] — Adjusted gMean ratio of test/reference (T/R). Intra-individual geometric coefficient of variation (gCV) = 23.9%

2. Primary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Cmax)
Description: Maximum measured concentration of midazolam in plasma (Cmax).
  Detailed timeframe: For midazolam (R): Within 3 hours prior to midazolam administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after midazolam administration in period 1. For BI + midazolam (T): 313 hours prior to administration of BI 1015550 + midazolam, at BI 1015550 + midazolam administration (0 hour) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after administration of BI 1015550 + midazolam in period 2.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomol per Liter (nmol/L)
Groups:
- BI 1015550 + Midazolam (T): One film-coated tablet of 18 mg BI 1015550 was administered orally twice daily (bid) on Days -13 to -1, and once daily (qd) on Day 1 together with a single dose of 1 mL oral solution of midazolam (2mg/mL) as test treatment (T) in period 2.
Arm/Group | Midazolam (R) | BI 1015550 + Midazolam (T)
Number analyzed (Participants) | 15 | 15
Nanomol per Liter (nmol/L) | 28.0 (NA) — Adjusted geometric standard error (gSE) = 1.082 | 21.8 (NA) — Adjusted geometric standard error (gSE) = 1.082
Statistical Analysis 1: Comparison: Midazolam (R) vs BI 1015550 + Midazolam (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; adjusted gmean Ratio (%) = 78.0, 90% CI 2-sided [68.9 to 88.2] — Adjusted gMean ratio of test/reference (T/R). Intra-individual geometric coefficient of variation (gCV) = 19.4%

3. Secondary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of midazolam in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Detailed timeframe: For midazolam (R): Within 3 hours prior to midazolam administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after midazolam administration in period 1. For BI + midazolam (T): 313 hours prior to administration of BI 1015550 + midazolam, at BI 1015550 + midazolam administration (0 hour) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after administration of BI 1015550 + midazolam in period 2.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Hours * nanomol per liter (h*nmol/L)
Arm/Group | Midazolam (R) | BI 1015550 + Midazolam (T)
Number analyzed (Participants) | 15 | 15
Hours * nanomol per liter (h*nmol/L) | 80.8 (NA) — Adjusted geometric standard error (gSE) = 1.115 | 72.6 (NA) — Adjusted geometric standard error (gSE) = 1.115
Statistical Analysis 1: Comparison: Midazolam (R) vs BI 1015550 + Midazolam (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; adjusted gmean Ratio (%) = 89.8, 90% CI 2-sided [76.9 to 104.9] — Adjusted gMean ratio of test/reference (T/R). Intra-individual geometric coefficient of variation (gCV) = 24.4

ADVERSE EVENTS:
Time Frame: For Midazolam: At midazolam administration, plus 12 hours of residual effect period (REP), up to 12 hours. For BI 101550 and BI 101550 + Midazolam: From first drug administration until last drug administration, plus REP of 7 days, up to 21 days.
Description: Treated Set (TS): This set included all subjects who were treated with at least 1 dose of trial drug.
Groups:
- Midazolam: A single dose of 1 mL of midazolam solution (2mg/mL) was administered orally on Day 1 as reference treatment (R ) in period 1.
- BI 1015550: One film-coated tablet of 18 mg BI 1015550 was administered orally twice daily (bid) for 13 days (Day -13 to Day -1), and once daily (qd) on Day 1 in period 2.
- BI 101550 + Midazolam: One film-coated tablet of 18 mg BI 1015550 was administered orally twice daily (bid) for 13 days (Day -13 to Day -1), and once daily (qd) on Day 1 together with a single dose of 1 mL oral solution of midazolam (2mg/mL) as test treatment (T) in period 2.
Arm/Group | Midazolam | BI 1015550 | BI 101550 + Midazolam
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 9/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam (N=15) | BI 1015550 (N=15) | BI 101550 + Midazolam (N=15)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 0 | 2 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review Prior to any Submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI´s intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT05550636/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT05550636/SAP_001.pdf